CLINICAL TRIAL: NCT04877743
Title: A Phase IV Non-Interventional Enhanced Active Surveillance Study of Adults Vaccinated With AZD1222
Brief Title: Non-Interventional Enhanced Active Surveillance Study of Adults Vaccinated With AZD1222
Acronym: COVID-19
Status: Terminated | Type: Observational
Why Stopped: The AZ:CONNECTEU study will be stopped. Ongoing participants will be informed and off-boarded. Vaxzevria's safety continues to be monitored through the implementation of other studies and through established safety reporting platforms across Europe.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111R00003
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Active Surveillance Study; Non-interventional; Post-authorisation safety studies; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: This prospective cohort study will include participants who receive the AZD1222 vaccine. Enrolment is permitted within 28 days of the first dose of AZD1222 and can be completed at the vaccination site or remotely.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — The main data sources for the study will be participants and their medical records. Vaccination details will be verified by a vaccination card, batch/lot number, and/or using a regional vaccination register. Participants will report all study outcomes using the study app, web portal, or call centre. Participants can also select a proxy to communicate on their behalf: a caregiver, family member, or other trusted individual. Participants will be asked for an emergency contact in case of death or incapacity.

SUMMARY:
This is a Phase IV real-world, observational, non-interventional, prospective cohort study of adults vaccinated with AZD1222. The purpose of this study is to assess the safety and tolerability of AZD1222 in adults vaccinated in real-world settings.

DETAILED DESCRIPTION:
The study will use an innovative digital platform (study app and web portal) as well as a traditional call centre to collect participant responses to a series of health and well-being questionnaires over an 18-month period.

Research coordinators at vaccination sites will invite vaccinated adults to join the study. Participants can enrol at the vaccination site with assistance from a research coordinator or can take home a study information brochure and enrol within 28 days after the first dose of AZD1222. Research coordinators and the study call centre will be available to assist with enrolment and informed consent, as needed. Electronic consent using the study app will be an option where permitted.

Participants using the digital platform will set up a secure account, complete the enrolment questionnaires, and provide details of their vaccination to confirm eligibility. Non-digital participants will complete the enrolment questionnaires and confirm eligibility at a vaccination site or by a telephone call to the call centre. After enrolment, participants will be contacted to complete follow-up questionnaires at timed intervals over an 18-month period after their first AZD1222 dose. Digital participants will receive push notifications or emails and non-digital participants will receive phone calls. Participants can also submit unscheduled adverse event (AE) reports through the digital platform and call centre.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older at the time of vaccination.
* Received AZD1222 as the first dose of COVID-19 vaccination in the prior 28 days.
* The participant has provided sufficient details to validate the vaccination (vaccination card, batch/lot number, and/or regional vaccination register details).
* Provided informed consent to participate in the study, either personally or through a legal representative.
* Able and willing to provide responses to study notifications using the mobile device app, web portal, or call centre or have a proxy (a caregiver, family member, or other trusted individual) who can do so on their behalf.
* Able and willing to grant, personally or through a legal representative, permission to contact the participant's healthcare providers and to access the participant's medical records at the time of vaccination and during the post-vaccination follow-up period.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be adults ≥ 18 years of age who receive the AZD1222 vaccine in Germany, France, Spain, or Sweden and are able and willing to consent to participate in the study. This study will enrol all eligible participants but, in particular, will seek to enrol older adults, with a target of 50% of participants being aged ≥ 65 years. Other subpopulations of interest include pregnant women, women who are breastfeeding, immunocompromised persons, persons with an autoimmune or inflammatory disorder, and frail persons with comorbidities. The study will also aim for an approximately equal enrolment of male and female participants.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAEs), adverse events of special interest (AESIs) and medically-attended adverse events following immunisation (AEFIs) with AZD1222 for 3 months after vaccination | Up to 3 months
  The incidence of SAEs, AESIs, and medically-attended AEFIs after at least one intramuscular (IM) dose of AZD1222 will be estimated for 3 months after vaccination.

SECONDARY OUTCOMES:
Number of participants with SAEs, AESIs and medically-attended AEFIs with AZD1222 for up to 18 months after vaccination | Up to 18 months
  The incidence of SAEs, AESIs, and medically-attended AEFIs after at least one IM dose of AZD1222 will be estimated for up to 18 months after vaccination.
Number of participants with SAEs, AESIs and medically-attended AEFIs with AZD1222 categorised by age group | Up to 18 months
  The incidence of SAEs, AESIs, and medically-attended AEFIs after at least one IM dose of AZD1222 will be estimated in participants by age group.
Number of participants with select comorbidities with SAEs, AESIs and medically-attended AEFIs with AZD1222 | Up to 18 months
  The incidence of SAEs, AESIs, and medically-attended AEFIs after at least one IM dose of AZD1222 will be estimated in participants with select comorbidities.
Prevalence of pregnancies resulting in spontaneous abortions within the AESI medical concept of Pregnancy Outcomes - Maternal | Up to 12 months
  The frequency of select pregnancy outcomes will be estimated in women vaccinated with AZD1222 during pregnancy or within 45 days of the estimated conception date.
Prevalence of pregnancies resulting in stillbirths within the AESI medical concept of Pregnancy Outcomes - Maternal | Up to 12 months
  The frequency of select pregnancy outcomes will be estimated in women vaccinated with AZD1222 during pregnancy or within 45 days of the estimated conception date.
Prevalence of pregnancies resulting in preterm births within the AESI medical concept of Pregnancy Outcomes - Maternal | Up to 12 months
  The frequency of select pregnancy outcomes will be estimated in women vaccinated with AZD1222 during pregnancy or within 45 days of the estimated conception date.
Prevalence of major congenital malformations in the AESI medical concept of Pregnancy Outcomes - Neonates as a measure of infant outcome | Up to 12 months
  The frequency of select outcomes will be estimated at birth and up to 12 months of age in neonates/infants born to mothers vaccinated with AZD1222 during pregnancy or within 45 days of the estimated conception date.
Prevalence of small for gestational age in the AESI medical concept of Pregnancy Outcomes - Neonates as a measure of infant outcome | Up to 12 months
  The frequency of select outcomes will be estimated at birth and up to 12 months of age in neonates/infants born to mothers vaccinated with AZD1222 during pregnancy or within 45 days of the estimated conception date.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00003&attachmentIdentifier=8ebea781-8100-44d5-89bc-6427d93bb32a&fileName=d8111r00003_(Pxl_257664)-clinical-study-report_Abstract__Redacted.pdf&versionIdentifier=